CLINICAL TRIAL: NCT06007456
Title: Clinical, Laboratory and Ultrasound Stratification of Patients With Juvenile Idiopathic Arthritis and Outcomes Evaluation During Transition to Adult Care
Brief Title: Clinical, Laboratory and Ultrasound Stratification of Patients With Juvenile Idiopathic Arthritis
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 23/22
Record Dates: First submitted 2023-03-28; First posted 2023-08-23 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: JIA; classification; transition of care
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients at onset of juvenile arthritis: New diagnosis of JIA
- Patients with juvenile arthritis in follow up: Subjects with JIA already followed at Rheumatologic Service

SUMMARY:
Juvenile Idiopathic Arthritis (JIA), the most common rheumatologic chronic disease in children, is defined as arthritis persisting for at least 6 weeks with no known cause in a patient under the age of 16. The term JIA is an umbrella that includes very different diseases. The current International League of Associations for Rheumatology (ILAR) classification divides JIA patients into 7 categories based on number of involved joints and time of involvement, presence of systemic symptoms, psoriatic findings and spondyloarthritis. This classification groups together patients with different disease and divides patients with the same disease. In the first case, unifying distinct diseases could lead to undifferentiated therapeutic choices, moving away from the modern concept of therapeutic personalization. In the second case, similarities between paediatric and adult arthritis could not be found. This involves both a loss of collaboration with the adult rheumatologist and the difficulty in accessing possibly effective therapies approved only for adult arthritis.

In clinical practice, it is increasingly evident that the number of affected joints and the speed of joint involvement are not useful criteria for defining the type and severity of disease. Joint counts lead to underestimate the importance of joint distribution in the identification of distinct forms of arthritis. A recent study found that patterns of joint involvement represent prognostic features, so grouping patients by joint pattern and degree of localization may help clinicians tailor treatments based on predicted disease trajectories. Another important point to differentiate some forms of arthritis is the presence of enthesitis and tenosynovitis. Sometimes tendon inflammation can be not clinically evident, so ultrasound evaluation is useful to detect it. Musculoskeletal ultrasound (MSUS) has been used worldwide by adult rheumatologist, but it is beginning a useful tool also in patients with JIA. Recent studies underline the important role of MSUS findings to assess disease activity and assist disease classification. In recent years, the need has emerged to replace the ILAR criteria with a new nomenclature based on the disease biology. This approach could help clinicians to choose a personalized therapeutic strategy for patients with arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects under the age of 18 years
* Arthritis persisting for at least 6 weeks with no known cause

Exclusion Criteria:

* No consent from the patients' guardians
* Patients with Systemic onset Juvenile Idiopathic Arthritis
* Patients who developed arthritis on a pre-existing inflammatory disorder such as Inflammatory Bowel Disease, and had received previous treatments

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with JIA during the transition to adult care
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate disease activity by the Juvenile Arthritis Disease score during the transition to adult care | Between 14-17 years of age
  The Juvenile Arthritis Disease score (JADAS) includes 4 measures: physician's global assessment of disease activity, measured on a 0-10 visual analog scale (VAS) (0=no activity-10=maximum activity); parent global assessment of well-being, measured on a 0-10 VAS (0=very well-10=very poor); the erythrocyte sedimentation rate, normalized to a 0 to 10 scale; and a count of joints with active disease. The final score is calculated as the sum of the scores of these four components (higher scores indicate higher disease activity).
To evaluate disease activity by the Health Assessment Questionnaire - Disability Index during the transition to adult care | Between 14-17 years of age
  The Health Assessment Questionnaire - Disability Index (HAQ-DI) includes 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities, with 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section. The 8 scores of the 8 sections are summed and divided by 8.
To assess joint damage by radiological examination during the transition to adult care | Between 14-17 years of age
  Radiographs will be performed to assess the presence of joint damage

SECONDARY OUTCOMES:
To evaluate non-inflammatory pain by the widespread pain index scale during transition to adult care | Between 14-17 years of age
  Pain will be evaluated through the widespread pain index (WPI) scale that assesses the presence of pain in 19 designated body locations over the past 7 days. Each location is equal to a score of 1. The WPI indicates the total number of areas that are painful, giving a maximum value of 19. WPI score can range from 0 to 19.

CONTACTS AND LOCATIONS:
Overall Officials: Serena Pastore, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (2):
- Italy (2):
  - IRCCS Burlo Garofolo, Trieste
  - (Department of Medical and Biological Sciences, Rheumatology Clinic, University of Udine, Udine